CLINICAL TRIAL: NCT00781898
Title: Prevention of Relapse to Opioid Addiction Using Depot Naltrexone
Brief Title: Treatment Study Using Depot Naltrexone (1/6) Philadelphia Coord/Data Mgmt Site
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 808422; R01DA024553 (NIH)
Record Dates: First submitted 2008-10-24; First posted 2008-10-29 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Opiate Addiction
Keywords: Depot naltrexone; Parolees; Opioid addiction prevention; Medication Treatment Alternatives; Prevention of Relapse to Opioid Addiction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Depot Naltrexone (Active Comparator)
  Interventions: Drug: Depot naltrexone
- Placebo (Placebo Comparator)
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Drug: Depot naltrexone — Vivitrol® extended release naltrexone 380 mg per month delivered in monthly intramuscular injections.
  Arms: Depot Naltrexone
Other: Treatment as Usual (TAU) — Treatment as Usual (TAU) community treatment provided to the participant
  Arms: Placebo

SUMMARY:
The aim of this project is to conduct a multi-site effectiveness study to determine whether the addition of a monthly injection of depot naltrexone to treatment as usual (TAU) will significantly improve outcome in parolees and probationers with a history of opioid addiction compared to TAU alone. Participants will be randomized to either treatment as usual in community programs or monthly injections of depot naltrexone for six months with treatment as usual in community programs. The effectiveness of depot naltrexone has never been studied in opioid dependent parolees. all parolee subjects will be evaluated at baseline, while in treatment, and at 6, 12 and 18 month post entry time points. The primary study outcomes are retention in treatment, drug use, re-arrests, psychosocial and medical/psychiatric functioning, and economic costs and benefit costs of naltrexone.

DETAILED DESCRIPTION:
This site serves as the coordinating center for five sites conducting the trial under the same IND and same protocol.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 60;
* Have dx of opioid dependence according to DSM-IV criteria
* be in good general health as determined by complete physical and laboratory tests;
* Under some form of criminal justice supervision for at least 12 months;
* Have a negative result for urinary opioids and no sign of opiate withdrawal after IV (or IM) injection of 0.8 mg of naloxone; and
* Express a goal of opiate free treatment rather than agonist maintenance

Exclusion Criteria:

* Current drug or alcohol dependence that requires medical supervision;
* untreated psychiatric disorders that might make participation hazardous (e.g. untreated psychosis, bipolar disorder with mania, significant suicide risk). Adequately treated psychiatric disorders and appropriate psychotropic medications would be allowed.

  3. Active medical illness that might make participation hazardous (e.g., untreated hypertension, hepatitis with AST or ALT >3 times upper limit of normal, unstable diabetes or heart disease). Adequately treated medical conditions are acceptable; 4. female subjects who are pregnant or lactating, or female subjects of childbearing potential who are not using birth control (oral contraceptives, barrier (diaphragm or condom) plus spermicide, or levonorgestriel implant); 5. Liver failure or liver function test levels greater than three times normal; 6. History of allergic reaction to naltrexone; 7. History of a drug overdose in the past 3 years; and 8. Current diagnosis of chronic pain disorder for which opioids are prescribed for pain relief.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2008-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles P O'Brien, MD, PhD, Principal Investigator — University of Pennsylvania; James W Cornish, MD, Principal Investigator — University of Pennsylvania; Donna Coviello, PhD, Principal Investigator — University of Pennsylvania; Peter Friedmann, MD, MPH, Principal Investigator — Rhode Island Hospital; Timothy Kinlock, PhD, Principal Investigator — Mountain Manor Treatment Center, Baltimore MD; Edward B. Nunes, MD, Principal Investigator — New York State Psychiatric Institute, New York, NY; Josh Lee, MD, Principal Investigator — New York University/Bellevue
Locations (1):
- Treatment Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Chen DT, Ko TM, Allen AA, Bonnie RJ, Suratt CE, Appelbaum PS, Nunes EV, Friedmann PD, Lee JD, Gordon MS, McDonald R, Wilson D, Boney TY, Murphy SM, O'Brien CP. Personal Control Over Decisions to Participate in Research by Persons With Histories of Both Substance Use Disorders and Criminal Justice Supervision. J Empir Res Hum Res Ethics. 2018 Apr;13(2):160-172. doi: 10.1177/1556264618755243. Epub 2018 Feb 20. PMID 29460668
- [Derived] Lee JD, Friedmann PD, Kinlock TW, Nunes EV, Boney TY, Hoskinson RA Jr, Wilson D, McDonald R, Rotrosen J, Gourevitch MN, Gordon M, Fishman M, Chen DT, Bonnie RJ, Cornish JW, Murphy SM, O'Brien CP. Extended-Release Naltrexone to Prevent Opioid Relapse in Criminal Justice Offenders. N Engl J Med. 2016 Mar 31;374(13):1232-42. doi: 10.1056/NEJMoa1505409. PMID 27028913
- [Derived] Lee JD, Friedmann PD, Boney TY, Hoskinson RA Jr, McDonald R, Gordon M, Fishman M, Chen DT, Bonnie RJ, Kinlock TW, Nunes EV, Cornish JW, O'Brien CP. Extended-release naltrexone to prevent relapse among opioid dependent, criminal justice system involved adults: rationale and design of a randomized controlled effectiveness trial. Contemp Clin Trials. 2015 Mar;41:110-7. doi: 10.1016/j.cct.2015.01.005. Epub 2015 Jan 17. PMID 25602580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community-dwelling adult volunteers who had been incarcerated and who had a history of opioid dependence.
Period: Overall Study
Arm/Group | Depot Naltrexone | Placebo
Started | 153 | 155
Completed | 119 | 126
Not Completed | 34 | 29

BASELINE CHARACTERISTICS:
Population: Participants in this arm were randomized to Depot Nalttrexone (Extended Release Naltrexone)
Groups:
- Depot Naltrexone: Participants who were randomized to receive Extended Release Naltrexone
- Total: Total of all reporting groups
Arm/Group | Depot Naltrexone | Placebo | Total
Number analyzed (Participants) | 153 | 155 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 153 | 155 | 308
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (9.2) | 43 (9.4) | 43.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 129 | 132 | 261
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 153 | 155 | 308

OUTCOME MEASURES:

1. Primary Outcome: Relapse
Description: A relapse event was defined as 10 or more days of opioid use in a 28-day (4-week) period as assessed by self-report or by testing of urine samples obtained every 2 weeks; a positive or missing sample was computed as 5 days of opioid use.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Depot Naltrexone | Placebo
Number analyzed (Participants) | 153 | 155
Participants | 66 | 99

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse Events were assessed at each study visit
Arm/Group | Depot Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 2/153 | 5/155
Serious Adverse Events (participants affected / at risk) | 16/153 | 45/155
Other Adverse Events (participants affected / at risk) | 29/153 | 13/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depot Naltrexone (N=153) | Placebo (N=155)
Depression or suicidality (Psychiatric disorders) | 3 | 6
Chest pain (Cardiac disorders) | 2 | 4
Death (General disorders) | 2 | 5
Musculoskeletal symptom (Musculoskeletal and connective tissue disorders) | 2 | 4
Stroke (Cardiac disorders) | 2 | 0
COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Abscess (Skin and subcutaneous tissue disorders) | 0 | 4
Nonfatal Overdose (General disorders) | 0 | 4
Exacerbation of Pre-existing condition (General disorders) | 0 | 3
Surgery for Colon Cancer (Surgical and medical procedures) | 0 | 2
Any Overdose (General disorders) | 0 | 7
Fatal Overdose (General disorders) | 0 | 3
Stroke (General disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Dehydration (General disorders) | 1 | 0
Acute Renal failure (Renal and urinary disorders) | 1 | 0
Opioid Withdrawal (General disorders) | 1 | 0
Hospitalization Unknown (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depot Naltrexone (N=153) | Placebo (N=155)
Headache (General disorders) | 29 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No